CLINICAL TRIAL: NCT04457973
Title: Home-based Transcranial Direct Current Stimulation (tDCS) for Pain Management in Persons With Alzheimer's Disease and Related Dementias
Brief Title: Home-based Transcranial Direct Current Stimulation for Pain Management in Persons With Alzheimer's Disease and Related Dementias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Hyochol Ahn, PhD, Associate Dean for Research & Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-SN-20-0640; R15NR018050 (NIH)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer's Disease and Related Dementias
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental)
  Interventions: Device: Active tDCS
- Sham tDCS (Placebo Comparator)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — tDCS with a constant current intensity of 2 milliampere (mA) will be applied for 20 minutes per session daily for 5 days via the Soterix 1x1 tDCS mini-CT Stimulator device with headgear and 5x7 cm saline-soaked surface sponge electrodes.
  Arms: Active tDCS
Device: Sham tDCS — The electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds.
  Arms: Sham tDCS

SUMMARY:
The purpose of this project is to evaluate the preliminary effects of home-based M1-SO applied tDCS (that is, tDCS with the anode over the primary motor cortex and the cathode over the contralateral supraorbital area) on clinical pain in persons with early-stage Alzheimer's disease and Related Dementias (ADRD), to evaluate the preliminary effects of home-based M1-SO applied tDCS on pain-related cortical response in persons with early-stage ADRD, and to evaluate the feasibility and acceptability of home-based M1-SO applied tDCS for pain management in persons with early-stage AD.

ELIGIBILITY:
Inclusion Criteria:

* early-stage Alzhimer's disease and related dementias (ADRD)
* have caregiver-reported chronic pain (average pain in the past 3 months ≥ 3 out of 10),
* have a caregiver willing to participate in the study who sees the participant at least 10 hours/week
* can speak and read English
* have no plans to change medication regimens during the trial

Exclusion Criteria:

* history of brain surgery, brain tumor, seizure, stroke, or intracranial metal implantation
* alcohol/substance abuse
* severely diminished cognitive function (i.e., MiniMental Status Exam score ≤ 15)
* hospitalization within the preceding year for neuropsychiatric illness

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyochol Ahn, RN,PhD,MSN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham tDCS: Sham tDCS: The electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds out of 20 minutes per session daily for 5 days via the Soterix 1x1 tDCS mini-CT Stimulator device with headgear and 5x7 cm saline-soaked surface sponge electrodes.
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active tDCS: 2mA current is applied for 20 minutes.
- Sham tDCS: 2mA current is applied for 30 seconds.
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.10 (6.20) | 71.90 (8.97) | 73 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain as Assessed by the Mobilization-Observation-Behavior-Intensity-Dementia (MOBID-2) Scale
Description: Mobilization-Observation-Behavior-Intensity-Dementia (MOBID-2) is a 10 question scale, each question rated from 0-10. The total score ranges between 0-100 with a higher number indicating a worse outcome. The change in total score between the baseline (day 1) and the end of intervention (day 5) is reported.
Time Frame: baseline (day 1), end of intervention (day 5)
Population: Comparison of pain intensity changes between two groups at 5 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
score on a scale | -2.70 (2.39) | -.40 (1.67)

2. Secondary Outcome: Clinical Pain as Assessed by a Numerical Rating Scale (NRS)
Description: Numeric Rating Scale (NRS) total score ranges from 0 (no pain) to 100 (most intense pain imaginable). The change in total score between the baseline (day 1) and the end of intervention (day 5) is reported.
Time Frame: baseline (day 1), end of intervention (day 5)
Population: Comparison of pain intensity changes between two groups at 5 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
score on a scale | -13.55 (14.90) | -3.30 (14.81)

3. Secondary Outcome: Behavioral and Psychological Symptoms of Dementia (BPSD) as Measured by the Cohen-Mansfield Agitation Inventory (CMAI)
Description: Cohen-Mansfield Agitation Inventory (CMAI) is a 29 question scale, each question measured from 1-7. Total score ranges from 29-203 with a higher score indicating a worse outcome. The change in total score between the baseline (day 1) and the end of intervention (day 5) is reported.
Time Frame: baseline (day 1), end of intervention (day 5)
Population: Comparison of CMAI score changes between two groups at 5 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
score on a scale | -2.35 (5.99) | -2.95 (5.24)

4. Secondary Outcome: Behavioral and Psychological Symptoms as Assessed by Neuropsychiatric Inventory (NPI)
Description: Neuropsychiatric Inventory (NPI) total score ranges from 0-144, with a higher score indicating greater symptoms. The change in total score between the baseline (day 1) and the end of intervention (day 5) is reported.
Time Frame: baseline (day 1), end of intervention (day 5)
Population: Comparison of NPI score changes between two groups at 5 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
score on a scale | -2.9 (15.08) | -2.30 (11.59)

5. Secondary Outcome: Change in Pain Related Cortical Response Using a Continuous Wave, Multichannel Functional Near-infrared Spectroscopy (fNIRS) Imaging System
Description: Pain-related cortical response will be measured during thermal pain stimulation using a continuous-wave, multichannel fNIRS imaging system (LIGHTNIRS, Shimadzu, Kyoto, Japan) composed of 8 source and 8 detector channels.
  fNIRS signals between each source-to-detector pair are analyzed using a general linear model, Y = X*Beta + E , to test for statistical differences between the baseline (day 1) and the end of intervention (day 5).
  Y is the measured fNIRS signal, X is an array encoding the expected/hypothetical response, E is an error term, and Beta is interpreted as the strength/amplitude of the functional activation.
  Greater absolute Beta values denote that the change in cortical response between two sessions is greater.
  The calculated Beta values are expressed in arbitrary units.
Time Frame: baseline (day 1), end of intervention (day 5)
Population: Comparison of Beta value changes between two groups at 5 days from baseline.
Measure: Number; unit: Beta value
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
Beta value
  source 1, detector 1 | -6.39 | -5.30
  source 2, detector 2 | 2.31 | -4.64
  source 3, detector 3 | -3.60 | 3.13
  source 4, detector 4 | -8.35 | -3.46
  source 5, detector 5 | -1.03 | -1.54
  source 6, detector 6 | -1.99 | -3.49
  source 7, detector 7 | -1.61 | -0.97
  source 8, detector 8 | 3.88 | 8.33

6. Secondary Outcome: Acceptability as Measured by the tDCs Experience Questionnaire
Description: The tDCS experience questionnaire contains 10 questions based on a scale from 0-10, 0 being strongly disagree and 10 being strongly agree. Higher scores indicating greater acceptability for 7 questions and lower scores indicating greater acceptability for 3 reversed questions. Total score ranges from 0-100 with a most desirable score of a 70.
Time Frame: end of intervention (day 5)
Population: Comparison of total score of tDCS experience questionnaire between two groups at 5 days from baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
score on a scale | 62.05 (8.76) | 67.95 (11.06)

7. Secondary Outcome: Patient Satisfaction as Measured by the Client Satisfaction Questionnaire (CSQ)
Description: Client Satisfaction Questionnaire (CSQ) consists of 8 questions, each is rated between 1-4. The total score ranges from 8-32 with a higher score indicating a higher satisfaction.
Time Frame: end of intervention (day 5)
Population: Comparison of total score of CSQ between two groups at 5 days from baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
score on a scale | 28.75 (2.92) | 28.55 (3.14)

ADVERSE EVENTS:
Time Frame: 1 week, from the first day of tDCS session to the last day.
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04457973/Prot_001.pdf
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04457973/SAP_002.pdf